CLINICAL TRIAL: NCT03733353
Title: A Phase 1 Randomized Double-Blind Placebo-controlled Single and Multiple Ascending Dose Study of EDP1815 in Healthy Participants and Participants With Mild to Moderate Psoriasis or Atopic Dermatitis
Brief Title: A Study of EDP1815 in Healthy Participants and Participants With Mild to Moderate Psoriasis and Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EDP1815-101; 2018-002807-32 (EudraCT Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Psoriasis; Atopic Dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: The study is a double-blind dose escalation cohort study in healthy volunteers and participants with either mild to moderate psoriasis or mild to moderate atopic dermatitis. The study consists of 10 cohorts and will test doses of EDP1815 versus placebo. The safety and tolerability of EDP1815 will be tested in participants with psoriasis and atopic dermatitis alongside pharmacodynamic effects on the systemic immune system and observation of any clinical effects.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1 (Other): 12 healthy volunteers; 8 on EDP1815, 4 on placebo. Dose=1/10th of HED, capsule, once daily, 15 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 2 (Other): 12 healthy volunteers; 8 on EDP1815, 4 on placebo. Dose= 1 x HED, capsule, once daily, 15 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 3 (Other): 12 subjects with mild to moderate psoriasis; 8 on EDP1815, 4 on placebo. Dose= 1 x HED, capsule, once daily, 29 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 4 (Other): 24 subjects with mild to moderate psoriasis; 16 on EDP1815, 8 on placebo. Dose= 5 x HED capsule, once daily, 29 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 5 (Other): 24 subjects with mild to moderate atopic dermatitis; 16 on EDP1815, 8 on placebo. Dose= 5 x HED, mini-tablets in capsule, once daily, 29 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 6 (Other): 24 subjects with mild to moderate psoriasis; 16 on EDP1815, 8 on placebo. Dose=5 x HED, mini-tablets in capsule, once daily, 29 days.
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 7 (Other): 24 subjects with mild to moderate atopic dermatitis; 16 on EDP1815, 8 on placebo. Dose= 5 x HED, capsule, once daily, 56 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 8 (Other): 24 subjects with mild to moderate psoriasis; 16 on EDP1815, 8 on placebo. Dose= 8 x HED, tablet, once daily, 56 days
  Interventions: Drug: EDP1815; Drug: Placebo oral tablet
- Cohort 9 (Other): 24 subjects with mild to moderate psoriasis; 16 on EDP1815, 8 on placebo. Dose= 2 x HED, capsule, once daily, 56 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule
- Cohort 10 (Other): 24 subjects with mild to moderate atopic dermatitis; 16 on EDP1815, 8 on placebo. Dose= 4 x HED, capsule, once daily, 56 days
  Interventions: Drug: EDP1815; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: EDP1815 — EDP1815 is an orally administered monoclonal microbial
Drug: Placebo oral capsule — Placebo
  Arms: Cohort 1; Cohort 10; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7; Cohort 9
Drug: Placebo oral tablet — Placebo
  Arms: Cohort 8

SUMMARY:
Evelo will investigate the safety and tolerability of EDP1815 and its potential to be a medicinal product in healthy volunteers and individuals with mild to moderate psoriasis and atopic dermatitis.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled clinical study with dose escalations to assess safety, tolerability, and pharmacodynamic effect of EDP1815. Since this clinical study is the first study in humans, the participants will be healthy volunteers or subjects with mild to moderate psoriasis or atopic dermatitis who are otherwise well. Investigation of EDP1815 in this patient population provides an opportunity to gain pharmacodynamic information using a range of tissue biopsies and composite clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

General:

Participant has a body mass index of ≥ 18 kg/m2 to ≤ 35 kg/m2 at Screening.

Healthy Volunteers:

Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.

Mild to moderate psoriasis:

1. Participant has had a confirmed diagnosis of mild to moderate plaque-type psoriasis for at least 6 months involving ≤ 10% of body surface area (BSA) (excluding the scalp).
2. Participant has a minimum of 2 psoriatic lesions with at least 1 plaque in a site suitable for biopsy.

Mild to moderate atopic dermatitis:

1. Mild to moderate atopic dermatitis with a minimum of 3% to a maximum of 15% BSA involvement.
2. Participant has had a confirmed diagnosis of mild to moderate atopic dermatitis for at least 6 months (IGA score of 2 or 3).
3. Participant has a minimum of 2 atopic dermatitis lesions with at least 1 in a site suitable for biopsy.

Exclusion Criteria:

1. Female participant who is pregnant, or plans to become pregnant during the study, or breastfeeding, or sexually active with childbearing potential who is not using a medically accepted birth control method.
2. Participant has received live attenuated vaccination within 6 weeks prior to Screening or intends to have such a vaccination during the course of the study.
3. Participant has received any investigational drug or experimental procedure within 90 days or 5 half-lives, whichever is longer, prior to study intervention administration.
4. Participant requires treatment with an anti-inflammatory drug during the study period. Paracetamol will be permitted for use as an antipyretic and/or analgesic (maximum of 4 grams/day in any 24 hour period).
5. Participant has an active infection (e.g. sepsis, pneumonia, abscess) or has had an infection requiring antibiotic treatment within 6 weeks prior to Investigational Medicinal Product (IMP) administration. When in doubt, the investigator should confer with the Sponsor study physician.
6. Participant has renal or liver impairment, defined as:

   1. For healthy volunteers: i. For women, serum creatinine level ≥ 125 μmol/L; for men, ≥ 135 μmol/L, or ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 1.5 x upper limit of normal (ULN), or iii. Alkaline phosphatase (ALP) and/or bilirubin > 1.5 x ULN
   2. For participants with mild to moderate atopic dermatitis or psoriasis: i. For women, serum creatinine level ≥ 125 μmol/L; for men, ≥ 135 μmol/L, or ii. ALT or AST > 2 x ULN and/or bilirubin > 1.5 x ULN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured through Adverse Events (AEs) | Day 1 to Day 70
  Number of participants with AEs by seriousness and relationship to treatment
Safety and tolerability measured through lab measurements | Day 0 to Day 70
  Number of participants with clinically significant change from baseline (Day 0) in laboratory values
Safety and tolerability measured through ECG | Day 0 to Day 70
  Number of participants with clinically relevant changes from baseline (Day 0) ECG parameters
Safety and tolerability measured through physical examination | Day 0 to Day 60
  Physical examination of stool samples based on the Bristol Stool Scale (Types 3 and 4 are ideal stool):
  Type 1: Separate hard lumps, like nuts (hard to pass); Type 2: Sausage-shaped, but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft; Type 5: Soft blobs with clear cut edges (easy to pass); Type 6: Fluffy pieces with ragged edges, a mushy stool; Type 7: Watery, no solid pieces, entirely liquid
GI safety measurement through biomarker analysis | Day 0 to Day 60
  GI safety measurement through fecal calprotectin analysis

SECONDARY OUTCOMES:
Clinical improvement in subjects with mild to moderate psoriasis | Day 0 to Day 70
  Change from baseline (Day 0) Psoriasis-area-and-severity index score (PASI) in response to EDP1815, measured on a scale of 0 to 6 (where 0 is most favorable and 6 is least favorable).
Clinical improvement in subjects with mild to moderate atopic dermatitis | Day 0 to Day 70
  Change from baseline (Day 0) Eczema-area-and-severity index score (EASI) in response to EDP1815, measured on a scale of 0 to 6 (where 0 is most favorable and 6 is least favorable).

CONTACTS AND LOCATIONS:
Overall Officials: Duncan McHale, MD, PhD, Study Director — Evelo Biosciences, Inc.
Locations (9):
- United Kingdom (9):
  - UK-8, Barnsley
  - UK-7, Blackpool
  - UK-3, Cannock
  - UK-4, Leeds
  - UK-5, Liverpool
  - UK-1, London
  - UK-2, Manchester
  - UK-6, Manchester
  - UK-9, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Itano A, Maslin D, Ramani K, Mehraei G, Carpenter N, Cormack T, Saghari M, Moerland M, Troy E, Caffry W, Wardwell-Scott L, Abel S, McHale D, Bodmer M. Clinical translation of anti-inflammatory effects of Prevotella histicola in Th1, Th2, and Th17 inflammation. Front Med (Lausanne). 2023 May 5;10:1070433. doi: 10.3389/fmed.2023.1070433. eCollection 2023. PMID 37215725